CLINICAL TRIAL: NCT06595173
Title: Therapeutic Artistic Activities in Adolescent with Diabetes
Brief Title: Effects of Therapeutic Artistic Activities on the Mental Status of Adolescents Followed Up with Diabetes Diagnosis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Çiğdem Sarı Öztürk, Gazi University, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSOZTURK/23-24
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Adolescent; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Theraputic Artistic activities group (Experimental): The group receiving therapeutic artistic activities
  Interventions: Behavioral: Therapeutic Intervention
- Standardized Control Group (No Intervention): the group that did not receive any training

INTERVENTIONS:
Behavioral: Therapeutic Intervention — group where therapeutic art activities such as mandala, drawing, third person singular method are applied.
  Therapeutic artistic activities within the program (drawing, zentagle, etc.). The program will be implemented in 6 weeks. At the beginning and end of the program, children's anxiety and psychological well-being levels will be evaluated.
  Arms: Theraputic Artistic activities group

SUMMARY:
This study will examine the effectiveness of therapeutic artistic activities in diabetic adolescents between the ages of 9-18. The study includes a 6-week program. The program will use art activities that can affect well-being, such as drawing a picture called a mandala. The State Anxiety Inventory will be used to measure the anxiety levels of adolescents, the Psychological Well-being Scale to assess their well-being, and a process evaluation form to evaluate the program (such as satisfaction).

DETAILED DESCRIPTION:
This study will be conducted with adolescents between the ages of 9-18 who are diagnosed with Type 1 Diabetes. The study includes a 6-week program. Art activities that can affect well-being, such as drawing a picture called a mandala, will be used in the program. Mandala drawing and painting will be done with the adolescents in the second and fourth weeks of the study. The drawings will be discussed in the third and fifth weeks. A common storytelling technique will be used according to the adolescents; feelings about drawing and painting. In the study, the State Anxiety Inventory will be used to measure the anxiety levels of the adolescents, the Psychological Well-being Scale to evaluate their well-being, and the process evaluation form where they evaluate the program (such as satisfaction). In addition, the Descriptive Characteristics Form, which consists of questions such as age and grade, will be applied in the first week of the study.

ELIGIBILITY:
Inclusion Criteria:

Adolescents who agree to participate in the study and whose parents give written consent,

* Are between the ages of 9-18,
* Have been diagnosed with Type 1 Diabetes at least 6 months ago,
* Have internet access on their smartphone or computer,
* Have no other physiological or psychological illness,
* Do not use psychoactive drugs

Exclusion Criteria:

* Those who use insulin pumps,
* Those who have experienced a significant life event in the last 6 months (such as migration, death, divorce in the family)
* Those who have practiced another body-mind based practice in the last 6 months (such as yoga, guided imagery, etc.)
* Those who do not have internet access

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Spielberger State Anxiety Inventory | Change from Baseline level of Spielberger State-Trait Anxiety to 5 weeks (change is being assessed)
  The scale is a 20-item self-report measure of anxiety using a 4-point Likert-type scale (from 0 to 3 points) for each item. The total score obtained from the scale varies between 20 and 60. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.
Psychological Well-Being Scale | Change from Baseline level of Adolescent Spiritual Well-Being Scale to 5 weeks (change is being assessed)
  The well-being scale developed by Diener and his colleagues was translated into Turkish by Telef (2013). The Psychological Well-being Scale consists of 8 items. The items of the scale are scored from strongly disagree (1) to strongly agree (7). The scores to be obtained from the scale vary between 8 and 56. The Cronbach alpha coefficient of the scale was calculated as 80.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gocen O, Ozturk CS. The effect of therapeutic artistic activities on anxiety and psychological well-being in adolescents with type 1 diabetes: a randomized controlled study. Eur J Pediatr. 2025 Jun 3;184(7):386. doi: 10.1007/s00431-025-06237-y. PMID 40461873